CLINICAL TRIAL: NCT00782080
Title: Efficacy and Safety of St. John´s Wort/Valerian Extract (Sedariston Concentrate) Versus Placebo in Children and Adolescents With Attention Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Efficacy and Safety of St. John´s Wort/Valerian Extract Versus Placebo in Children and Adolescents With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prof. Huss (Other)
Collaborators: Steiner Arzneimittel, Berlin, Germany (Unknown)
Responsible Party: Sponsor-Investigator, Prof. Huss, Prof. Dr. med. Dipl.-Psych. Michael Huss, Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Stei-Sed-0106
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: ADHD
Keywords: ADHD; children; adolescents; St. John's Wort; Valerian extract; Safety; Efficacy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sedariston (Experimental): Sedariston (100 mg St. John´s Wort and 50 mg Valerian extract) capsule given orally in capsules (size 1) twice daily for eight weeks in children (6-11): 1 - 0 -1 In Adolescents (12-17 years) two capsules (size 1) twice daily: 2 - 0 - 2.
  Interventions: Drug: Sedariston
- Placebo campsule (Placebo Comparator): Placebo provided by the company given orally in capsules (size 1 )twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sedariston — St. John´s Wort (100 mg) Valerian Extract (50 mg)
  Other Names: Sedariston Concentrate(R)
  Arms: Sedariston
Drug: Placebo — Placebo
  Arms: Placebo campsule

SUMMARY:
This study will determine the safety and efficacy of an herbal treatment in children and adolescents with ADHD.

Study Design:

* Randomized
* Double Blind (Subject, Caregiver, Investigator, Outcomes Assessor)
* Placebo Control
* Parallel Assignment

DETAILED DESCRIPTION:
ADHD is a common childhood disorder associated with attention problems and disruptive behavior. Clinical evidence suggests that a herbal drug combination of St. John´s Wort /Valerian extract may be effective in treating ADHD symptoms in methylphenidate and atomoxetine naive patients. This study will determine the safety and efficacy of an herbal treatment in children and adolescents with ADHD.

Participants will be randomly assigned to receive either an herbal product or placebo twice a day for the duration of 8 weeks. Participants will come in for study visits after 2 and 8 weeks for the assessment of ADHD symptoms, performance and spontaneous movements. Side effects will be monitored continuously and also assessed by rating scales.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Diagnosis of ADHD
* Score of ADHDRS-IV-Parent Version ≥24
* Sufficient knowledge of the German language
* Written Informed Consent by parents and patients
* Ability to swallow study medication
* Sexually mature and active adolescents with highly effective methods of birth control:

  * contraception according to Pearl-Index < 1
  * when use of oral contraceptives, additional methods of contraception (e.g. condoms) are necessary, i.e. double-barrier

Exclusion Criteria:

* Known hypersensitivity against St. John´s wort or Valerian root or one of the excipients
* Known hypersensitivity of the skin when exposed to sunlight
* All serious internal diseases, and for this reason: Current intake of the following medication:

  * Ciclosporin, Tacrolimus, Indinavir and other protease inhibitors in the anti-HIV treatment
  * Irinotecan and other cytostatics
  * anticoagulants of the Cumarin-type, Digoxin, Amitriptylin, Nortriptyline
  * Midazolam, Theophylline or other medication with photosensitive effects
* All severe psychiatric diseases except oppositional defiant disorders (according to items 21-28 SNAP-IV) and conduct disorders (according to items 41-45 SNAP-IV), and for this reason current intake of the following medication: antidepressants and other psychotropic medication
* Indication for hospitalization
* Suicidality (including suicidal thoughts): Score ≥3 in item 10 of MADRS
* Pregnancy, lactation
* IQ < 70
* Positive screening for metabolites of illegal drugs in urine
* Previous medication with stimulants and/or atomoxetine
* Psychotropic co-medication
* Placement in an institution on official or judicial ruling
* Parallel participation in another clinical trial according to German Drug Law (AMG), or less than 4 weeks ago
* Patients requiring a primary medication with methylphenidate during the study period of 8 weeks

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 155 (Actual)
Dates: Start 2008-07; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
ADHD-IV rating scale | Difference in total score between baseline and end of study

SECONDARY OUTCOMES:
Barkley´s Side Effects Rating Scale | Difference between baseline and each visit

CONTACTS AND LOCATIONS:
Overall Officials: Michael Huss, Prof. Dr., Principal Investigator — Johannes Gutenberg University, Mainz, Dep. of Child and Adolescent Psychiatry
Locations (5):
- Germany (5):
  - Rheinhessenfachklinik, Alzey
  - DRK Fachklinik für Kinder- und Jugendpsychiatrie, Bad Neuenahr
  - Praxis für Kinder- und Jugendpsychiatrie, Berlin
  - Charité University, Berlin
  - Johannes Gutenberg University, Mainz